CLINICAL TRIAL: NCT04542226
Title: Open Observational Study of Efficacy and Safety of Polyoxidonium in Complex Therapy of Hospitalized Patients With COVID-19
Brief Title: Observational Open Study of Polyoxidonium in Hospitalized Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Other Study IDs: Covid_v_1.0
Record Dates: First submitted 2020-09-08; First posted 2020-09-09 (Actual); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Infections, Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — azoximer bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients hospitalized with COVID-19: Patients eligible for enrollment into the study
  Interventions: Drug: Polyoxidonium

INTERVENTIONS:
Drug: Polyoxidonium — Polyoxidonium (azoximer bromide) is administered in the dose of 12 mg (contents of 2 vials) once daily intravenously (IV) for 3 days, then every other day intramuscularly (IM) on days 5-17 (the total treatment course is 10 injections)
  Other Names: azoximer bromide

SUMMARY:
The study is designed as an open observational non-comparative study of Polyoxidonium®, lyophilizate for solution for injections and topical application, 12 mg in hospitalized patients with coronavirus disease (COVID-19).

DETAILED DESCRIPTION:
The study was planned as an observation of Polyoxidonium® administered in addition to Russian Ministry of Healthcare (MoH) guidance for standard COVID-19 treatment. Regimens have no limitations to the use of concomitant therapy. The aim of the study is to observe the safety and efficacy of Polyoxidonium®, lyophilizate for solution for injections, 12 mg in addition to complex treatment of hospitalized patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. The hospitalized patient was administered Polyoxidonium, according to the instruction for medical usage in complex with Russian MoH guidance for treatment of COVID-19.
2. Verified coronavirus disease COVID-19, and at least one of the following:

   * severe disease: mechanical ventilation or oxygen supply required with blood oxygen saturation (SpO2) ≤ 94% on room air or tachypnea, respiratory rate ≥ 24 breaths per minute,
   * mild-moderate disease: SpO2 > 94% on room air or respiratory rate < 24 breaths per minute.
3. The patient signed an Informed Consent form for participation in this study.
4. The patient can understand all protocol requirements, perform the study procedures, and agree to all limitations specified in the protocol.
5. Male and female patients from 18 years of age.
6. Confirmed diagnosis of coronavirus disease (COVID-19): laboratory-confirmed Severe acute respiratory syndrome-related coronavirus 2 (SARS-CoV-2) infection as determined by polymerase chain reaction (PCR), or other commercial or public health assay in any specimen prior to inclusion.

Exclusion Criteria:

1. Pregnancy or breastfeeding.
2. Pathological condition that the study doctor considers significant enough to prevent enrolment of this patient.
3. Participation in any clinical study within 30 days before the Informed Consent form provided.
4. Hypersensitivity and/or intolerability to any ingredient of the investigational product.
5. Acute or chronic renal failure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients with verified diagnosis of COVID-19 administered Polyoxidonium, according to the instruction for its medical usage in complex with Russian MoH guidance for treatment of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay S. Dodonov, Study Chair — NPO Petrovax
Locations (5):
- Healthcare Institution "Grodno Regional Infectious Clinical Hospital", Grodno, Belarus
- Russia (4):
  - State-Funded Healthcare Institution "Emergency Hospital" of Ministry of Health of Chuvash Republic, Cheboksary, Chuvashskaya Respublika
  - State-Funded Healthcare Institution "Infectious Disease Hospital No.3" of Ministry of Health of Krasnodar Krai, Novorossiysk, Krasnodarskiy Kray
  - State-Funded Institution of Mari El Republic "Yoshkar-Ola City Hospital", Yoshkar-Ola, Mari El Republic
  - State-Funded Healthcare Institution of Voronezh Region "Novaya Usman District Hospital", Novaya Usman', Voronezh Oblast

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult Patients Hospitalized With COVID-19
Started | 81
Completed | 81
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.88 (12.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 77
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belarus | 10
  Russia | 71
Baseline severity according to the National Early Warning Score (NEWS Score) [Count of Participants; unit: Participants]
  Very Severe (NEWS ≥ 9) | 30
  Severe or Moderate (NEWS = 5…8) | 28
  Mild (NEWS ≤ 4) | 23
Respiratory support type [Count of Participants; unit: Participants]
  Invasive lung ventilation | 14
  Non-invasive lung ventilation | 25
  Oxygen therapy | 25
  None | 17
Mechanical ventilation [Count of Participants; unit: Participants]
  Present | 39
  Absent | 42
Basic concomitant medication [Count of Participants; unit: Participants]
  Antivirals | 46
  Antimalarial | 37
  Anticoagulants | 41
Ordinal Scale (OS) score [Mean (Standard Deviation); unit: units on a scale] — Clinical status assessment with 7-point ordinal scale (WHO Master Protocol [1])
  1. - Patient is not hospitalized, no limitations on activities;
  2. - Patient is not hospitalized, limitation on activities;
  3. - Patient is hospitalized, not requiring supplemental oxygen;
  4. - Patient is hospitalized, requiring supplemental oxygen;
  5. - Patient is hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. - Patient is hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO);
  7. - Death.
  units on a scale | 4.30 (1.02)
News Score (National Early Warning Score) [Mean (Standard Deviation); unit: units on a scale] — NEWS score is based on 7 clinical parameters:
  respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, temperature. A score of 0, 1, 2, 3 is allocated to each parameter except supplemental oxygen (a score 0 or 1 is allocated) and level of consciousness (a score 0 or 3 is allocated). A higher score means the parameter is further from the normal range. All scores were summed to get an aggregate score. Aggregate score ranges from 0 to 19, with higher scores meaning higher risk.
  units on a scale | 6.51 (3.41)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Status of the Patient (According to 7-point Ordinal Scale)
Description: Subject clinical status using the 7-point Ordinal Scale, specified as the primary endpoint in the WHO Master Protocol on day 15 as compared to baseline
  (1 - Not hospitalized, no limitations on activities; 2 - Not hospitalized, limitation on activities; 3 - Hospitalized, not requiring supplemental oxygen; 4 - Hospitalized, requiring supplemental oxygen; 5 - Hospitalized, on non-invasive ventilation or high flow oxygen devices; 6 - Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation; 7 - Death).
Time Frame: Day 1 (Baseline), Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Participants
  Number of patients at Baseline (Day 1): 1. Not hospitalized, no limitations on activities | 0
  Number of patients at Baseline (Day 1): 2. Not hospitalized, limitation on activities | 0
  Number of patients at Baseline (Day 1): 3. Hospitalized, not requiring supplemental oxygen | 22
  Number of patients at Baseline (Day 1): 4. Hospitalized, requiring supplemental oxygen | 24
  Number of patients at Baseline (Day 1): 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices | 24
  Number of patients at Baseline (Day 1): 6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation | 11
  Number of patients at Baseline (Day 1): 7. Death | 0
  Number of patients on Day 15: 1. Not hospitalized, no limitations on activities | 3
  Number of patients on Day 15: 2. Not hospitalized, limitation on activities | 27
  Number of patients on Day 15: 3. Hospitalized, not requiring supplemental oxygen | 37
  Number of patients on Day 15: 4. Hospitalized, requiring supplemental oxygen | 9
  Number of patients on Day 15: 5. Hospitalized, on non-invasive ventilation or high flow oxygen devices | 3
  Number of patients on Day 15: 6. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation | 2
  Number of patients on Day 15: 7. Death | 0
Statistical Analysis 1: Comparison: Adult Patients Hospitalized With COVID-19; Test type: Other; p < 0.0000001, Wilcoxon (Mann-Whitney) — the a priori threshold for statistical significance p<0.05; Wilcoxon signed-rank test for repeated measures was used to compare with baseline

2. Secondary Outcome: Time to Improvement in Clinical Status of the Patient (According to Ordinal Scale) by 1 Point for Each OS Score
Description: Ordinal scale (OS) score status, time to improvement by 1 point for each OS score.
  Subject clinical status using the 7-point Ordinal Scale:
  1. - Not hospitalized, no limitations on activities;
  2. - Not hospitalized, limitation on activities;
  3. - Hospitalized, not requiring supplemental oxygen;
  4. - Hospitalized, requiring supplemental oxygen;
  5. - Hospitalized, on non-invasive ventilation or high flow oxygen devices;
  6. - Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation;
  7. - Death.
Time Frame: Days 1 - 29.
Population: Administration of Polyoxidonium was canceled due to Adverse event in 1 patient. Patient received only 2 injections.This is the reason why the needed information for this Outcome Measure is absent for 1 patient.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 80
days | 13.77 (6.01)

3. Secondary Outcome: Clinical Status of the Patient (According to National Early Warning Score (NEWS Scale))
Description: NEWS scale score status, time to a discharge from a hospital or to a NEWS of ≤ 2 and maintained for 24 hours, whichever occurs first.
  NEWS score is based on 7 clinical parameters:
  respiration rate, oxygen saturation, supplemental oxygen, systolic blood pressure, pulse rate, level of consciousness, temperature. A score of 0, 1, 2, 3 is allocated to each parameter except supplemental oxygen (a score 0 or 1 is allocated) and level of consciousness (a score 0 or 3 is allocated). A higher score means the parameter is further from the normal range. All scores were summed to get an aggregate score. Aggregate score ranges from 0 to 19, with higher scores meaning higher risk.
  Low risk - aggregate score, 1-4 Low to medium risk - score 3 in any single parameter, Medium risk - aggregate score 5-6, High risk - aggregate score 7-19.
Time Frame: Days 1 - 29.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 80
days | 8.85 (6.10)

4. Secondary Outcome: Number of Patients Requiring Supplementary Oxygen
Description: Number of patients requiring supplementary oxygen on Days 3, 5, 8, 11, 15, 29
Time Frame: Days intervals 1 (baseline), 3, 5, 8, 11, 15, 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Participants
  Baseline (Day 1): Number of patients requiring supplementary oxygen | 59
  Baseline (Day 1): Number of patients not requiring respiratory support | 22
  Day 3: Number of patients requiring supplementary oxygen | 58
  Day 3: Number of patients not requiring respiratory support | 23
  Day 5: Number of patients requiring supplementary oxygen | 56
  Day 5: Number of patients not requiring respiratory support | 25
  Day 8: Number of patients requiring supplementary oxygen | 47
  Day 8: Number of patients not requiring respiratory support | 34
  Day 11: Number of patients requiring supplementary oxygen | 31
  Day 11: Number of patients not requiring respiratory support | 50
  Day 15: Number of patients requiring supplementary oxygen | 14
  Day 15: Number of patients not requiring respiratory support | 67
  Day 29: Number of patients requiring supplementary oxygen | 1
  Day 29: Number of patients not requiring respiratory support | 80

5. Secondary Outcome: Hospitalisation Duration
Description: Duration of hospitalisation
Time Frame: Days 1 - 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 80
days | 19.13 (5.29)

6. Secondary Outcome: Mortality
Description: Number of participants who were dead or alive (Days 1 - 29)
Time Frame: Days 1 - 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Participants
  Alive | 81
  Dead | 0

7. Secondary Outcome: The Number of Participants With Serious Adverse Events
Description: The number of participants with serious adverse events (SAE)
Time Frame: Days 1 - 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Participants | 1

8. Secondary Outcome: The Number of Participants With Adverse Events
Description: The number of participants with adverse events (AE)
Time Frame: Days 1 - 29.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Participants | 7

9. Secondary Outcome: Number of Participants With Discontinuation of Drug Administration
Description: Number of participants with Permanent or temporary discontinuation of infusions or injections due to adverse events
Time Frame: Days 1 - 17.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Patients Hospitalized With COVID-19
Number analyzed (Participants) | 81
Participants
  Administration of Polyoxidonium was canceled due to Adverse event | 1
  Administration of Polyoxidonium was postponed by 1 day due to Adverse event | 2

ADVERSE EVENTS:
Time Frame: Safety parameters were evaluated throughout the study in the Safety population (SAP; patients who received at least one Polyoxidonium dose, according to the prescribed treatment) from signing the informed consent to the study completion visit on Day 29±3.
Arm/Group | Adult Patients Hospitalized With COVID-19
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 1/81
Other Adverse Events (participants affected / at risk) | 6/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Patients Hospitalized With COVID-19 (N=81)
Klebsiella sepsis (Infections and infestations) | 1 (1) — This SAE was classified by the Investigator as not related to Polyoxidonium treatment. The patient had a history of previous bacterial pneumonias over the past 3 years.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Patients Hospitalized With COVID-19 (N=81)
PQ interval prolonged / Electrocardiogram PR prolongation* (Investigations) | 2 (2) — Patients received a combination of lopinavir+ritonavir, and this AEs was supposed by the Investigator to be caused by the antiviral drugs. After completion of antiviral treatment all symptoms eliminated and didn't require any additional actions.
Fever (Intermittent fever included) / Pyrexia (General disorders) | 3 (3) — Fever was apparently a result of SARS-CoV-2 infection and intoxication.It was classified by Investigators as not associated with Polyoxidonium treatment; some of them noted more rapid fever and intoxication decline in Polyoxidonium treated patients.
Pneumonia bacterial (Infections and infestations) | 1 (1) — Bacterial pneumonia was diagnosed. The Investigator did not associate the development of pneumonia with PO administration. Bacterial pneumonia is common COVID-19 complication in elderly patients.The investigator consider this event as AE.

LIMITATIONS AND CAVEATS:
There was no control or comparison group, polyoxidonium was used in the treatment of all patients, it is not possible to compare the results of treatment of patients with and without Polyoxidonium. The study used various treatment regimens for COVID-19 (antiviral agents, antimalarial agents, anticoagulants), depending on the base of the study, so it is impossible to fully determine whether these agents influenced the effectiveness of Polyoxidonium.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04542226/Prot_SAP_000.pdf